CLINICAL TRIAL: NCT05332691
Title: Minimally Invasive Transapical Septal Myectomy in the Beating Hearts for the Treatment of Hypertrophic Obstructive Cardiomyopathy: Safety and Efficacy Results of a Phase I First-in-man Clinical Trial
Brief Title: Transapical Beating-heart Septal Myectomy in Patient With Hypertrophic Obstructive Cardiomyopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiang Wei (Other)
Responsible Party: Sponsor-Investigator, Xiang Wei, Professor and Director, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-S013 2022-N016
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy
Keywords: Hypertrophic Obstructive Cardiomyopathy; Septal Myectomy; Systolic Anterior Motion; Left Ventricle Outflow Tract Obstruction; Mitral Regurgitation; Transapical; Off-pump; Minimally invasive
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Mitral Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Beating-heart myectomy device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypertrophic Obstructive Cardiomyopathy (Experimental): Transapical beating-heart septal myectomy for the patient with hypertrophic obstructive cardiomyopathy.
  Interventions: Procedure: Transapical beating-heart septal myectomy

INTERVENTIONS:
Procedure: Transapical beating-heart septal myectomy — We have invented a beating-heart myectomy device.Through a minimally invasive intercostal incision, septal myectomy could be accomplished via a transapical access in the beating heart using the device. The whole process of resection is monitored, navigated, and evaluated by real-time transesophageal and transthoracic echocardiography. Left ventricle outlet tract gradient and the grade of mitral regurgitation are evaluated each time after resection. Multiple resections are performed to tailor the muscular resection for sufficient relief of left ventricle outlet tract obstruction and mitral regurgitation, while preventing iatrogenic injuries.
  Other Names: Minimally invasive transapical septal myectomy in the beating hearts

SUMMARY:
The primary purpose of this study is to evaluate the feasibility, the safety and the efficacy of the transapical beating-heart septal myectomy for the treatment of hypertrophic obstructive cardiomyopathy. This is a prospective, single-arm, single-center, first-in-man study.

DETAILED DESCRIPTION:
Surgical septal myectomy remains the gold standard for the treatment of hypertrophic obstructive cardiomyopathy. However, conventional septal myectomy is hindered by the demanding expertise that is needed to sufficient relieve the obstruction of the left ventricle outflow tract while guarantee safety. To increase the visualization and minimize the surgical injury of conventional septal myectomy, we have invented a novel beating-heart myectomy device. Through a mini-thoractomy, septal myectomy could be accomplished via a transapical access in the beating heart using the beating-heart myectomy device. The whole process of resection is monitored, navigated, and evaluated by real-time transesophageal and transthoracic echocardiography. Left ventricle outflow tract gradient and the grade of mitral regurgitation are evaluated each time after resection. Multiple resections are performed to tailor sufficient relief of left ventricle outflow tract obstruction and mitral regurgitation, while preventing iatrogenic injuries. After transapical beating-heart septal myectomy, patients is scheduled to be seen for follow-up visits at discharge (about 7 days post operation) and 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose resting or provoked left ventricular outflow tract gradient > 50 mmHg, and maximal ventricular septal wall thickness ≥ 15 mm.
2. Patients with heart function of New York Heart Association ≥ class II.
3. Patients with drug-refractory symptoms or intolerable to pharmaceutical therapies.
4. Patients who was informed the nature of the clinical trial, consented to participate in all of the activities of the clinical trial, and signed the informed consent form.

Exclusion Criteria:

1. Patients who were pregnant.
2. Patients who had concomitant diseases such as intrinsic valvular disease or coronary artery disease that needed open-heart surgery.
3. Patients who had severe heart failure with left ventricle ejection fraction < 40%.
4. Patients whose estimated life expectancy < 12 m.
5. Patient who were non-compliant.
6. Patients under circumstances which were considered not suitable or prohibitive for participating the clinical trial at the discretion of the attending medical team and the researchers.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 3 months
  Death from any cause during the observation period.
Procedural success | 3 months
  Resting left ventricle outflow tract gradients < 30 mmHg, provoked left ventricle outflow tract gradients < 50 mmHg, and mitral regurgitation (MR) ≤ grade 1+.

SECONDARY OUTCOMES:
Device success | 1 day
  Successful accession, delivery, and retrieval of the resection device, successful resection of the septal myocardium, resting left ventricle outflow tract gradient less than 50 mmHg and mitral regurgitation (MR) ≤ grade 2+ during operation after resection, and free from conversion to midline thoracotomy during operation.
Septal thickness | 7 days and 3 months
  Basal and mid septal thickness as measured by echocardiography.
Left ventricle mass | 3 months
  Left ventricle mass index (the ratio of left ventricle mass to body weight) as measured by cardiac magnetic resonance.
Left ventricle volume | 7 days and 3 months
  Left ventricle end-diastolic volume as measured by echocardiography.
Cardiac diastolic function | 7 days and 3 months
  The ratio between early mitral inflow velocity and mitral annular early diastolic velocity ( E/e') as measured by echocardiography.
Left atria volume | 7 days and 3 months
  The left atria volume as measured by echocardiography.
Major adverse cardiovascular and cerebral events | 3 months
  In-hospital mortality, atrioventricular block that need permanent pacemaker implantation, sternotomy conversion, iatrogenic ventricular septal perforation, iatrogenic valvular injury, imaging examination-validated cerebral complications.
New York Heart Association class | 7 days and 3 months
  New York Heart Association class, including grade I, grade II, grade III, grade IV. A higher grade means worse heart function.
6-minute walking test | 3 months
  6-minute walking test. A longer distance means better heart function.
Heart function-associated quality of life | 7 days and 3 months
  Score of the Kansas City Cardiomyopathy Questionnaire. A higher score means better heart function.
Left ventricular outflow tract gradient | 7 days and 3 months
  Left ventricular outflow tract gradient as measured by echocardiography.
Evaluation of the mitral valve | 7 days and 3 months
  Grade of mitral regurgitation and systolic anterior motion as measured by echocardiography.
Left ventricular outflow tract diameter | 7 days and 3 months
  Left ventricular outflow tract diameter as measured by echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Wei, M.D., Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
All of the conclusive participant data, after removing the individual information of privacy, will be uploaded as supporting information when publishing the current study.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the current study is published.
Access Criteria: All readers who were interested in the current study.

REFERENCES:
- [Background] Fang J, Wang R, Liu H, Su Y, Chen J, Han X, Wei Y, Chen Y, Cheng L, Wei X. Transapical septal myectomy in the beating heart via a minimally invasive approach: a feasibility study in swine. Interact Cardiovasc Thorac Surg. 2020 Feb 1;30(2):303-311. doi: 10.1093/icvts/ivz249. PMID 31642911
- [Derived] Chen Y, Quintana E, Fang J, Liu Y, Wei X. Transapical Beating-Heart Septal Myectomy for Obstructive Hypertrophic Cardiomyopathy With Anomalous Papillary Muscle Insertion. Interdiscip Cardiovasc Thorac Surg. 2025 Sep 2;40(9):ivaf195. doi: 10.1093/icvts/ivaf195. PMID 40833749
- [Derived] Fang J, Chen Y, Liu Y, Li R, Zhu Y, Zhou W, Cheng L, Wang Q, Shi J, Wei Y, Ma Y, Quintana E, Grau JB, Wan S, Wei X. Transapical Beating-Heart Septal Myectomy for Obstructive Hypertrophic Cardiomyopathy: Lessons Learned After the Learning Curve Period. Circ Cardiovasc Interv. 2025 May;18(5):e015044. doi: 10.1161/CIRCINTERVENTIONS.124.015044. Epub 2025 May 2. PMID 40315478
- [Derived] Fang J, Liu Y, Zhu Y, Li R, Wang R, Wang DW, Song Y, Li C, Chen Y, Cheng L, Zheng K, Zhao Y, Li S, Cheng C, Xia L, Chen X, Wan S, Wei X. First-in-Human Transapical Beating-Heart Septal Myectomy in Patients With Hypertrophic Obstructive Cardiomyopathy. J Am Coll Cardiol. 2023 Aug 15;82(7):575-586. doi: 10.1016/j.jacc.2023.05.052. PMID 37558369

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT05332691/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT05332691/ICF_001.pdf